CLINICAL TRIAL: NCT03961191
Title: Utilization of DNA Methylation in the Screening of Uterine Cervical Lesions: A Case-control Study
Brief Title: DNA Methylation for Screening Uterine Cervical Lesions: A Case-control Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: METHY1
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: DNA Methylation; Uterine Cervical Cancer; High Grade Squamous Intraepithelial Lesions; Low Grade Squamous Intraepithelial Lesions
MeSH Terms: conditions — Uterine Cervical Neoplasms; Squamous Intraepithelial Lesions | interventions — DNA Methylation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Benign group: Patients with benign cervical histology, including normal findings, inflammation and LSIL
  Interventions: Diagnostic Test: DNA methylation; Diagnostic Test: high-risk HPV; Diagnostic Test: TCT
- HSIL group: Patients with cervical histology of HSIL
  Interventions: Diagnostic Test: DNA methylation; Diagnostic Test: high-risk HPV; Diagnostic Test: TCT
- Cancer group: Patients with cervical histology of cancer
  Interventions: Diagnostic Test: DNA methylation; Diagnostic Test: high-risk HPV; Diagnostic Test: TCT

INTERVENTIONS:
Diagnostic Test: DNA methylation — DNA methylation for the cervical cytology
Diagnostic Test: high-risk HPV — High-risk HPV testing for the cervical cytology
Diagnostic Test: TCT — Thin prep liquid-based cytology test for the cervical cytology

SUMMARY:
The primary objective of this study is to compare the testing of DNA methylation, high-risk HPV subtypes, and cytology with the definite histological results in a case-control study, so as to determine the accuracy of DNA methylation in the screening of uterine cervical lesions.

This study will include 300 patients with definite histological results, with 100 of cervical inflammation or low grade squamous intraepithelial lesions (LSIL), 100 of high grade squamous intraepithelial lesions (HSIL), and 100 of uterine cervical cancer. All the cervical specimens of cytology collected in the clinical settings will be utilized for the testing of DNA methylation, high-risk HPV subtypes and thin prep liquid-based cytology test (TCT). The sensitivity, specificity, positive predictive value and negative predictive value were calculated based on the known histological results. The differences of DNA methylation with high-risk human papillomavirus (HPV) and TCT will also be analyzed.

The testing of DNA methylation will be performed with the methylation-specific polymerase chain reaction (PCR). The TCT and HPV testing will be performed with the Roche kits.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cervical histology within one month when collecting cervical cytology
* Aged 18 years or older
* Signed an approved informed consents

Exclusion Criteria:

* Not meeting any of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Wtih confirmed cervical histology within one month when collecting cervical cytology
  2. Aged 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-05-22 (Actual); Primary Completion 2020-05-22 (Estimated); Study Completion 2020-05-22 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of DNA methylation | 1 years
  Sensitivity of DNA methylation compared with histological results for the differentiation of cervical cancer and HSIL
Specificity of DNA methylation | 1 years
  Specificity of DNA methylation compared with histological results for the differentiation of cervical cancer and HSIL

SECONDARY OUTCOMES:
Positive predictive value of DNA methylation | 1 year
  Positive predictive value of DNA methylation compared with histological results for the differentiation of cervical cancer and HSIL
Negative predictive value of DNA methylation | 1 year
  Negative predictive value of DNA methylation compared with histological results for the differentiation of cervical cancer and HSIL
Correlation coefficient of DNA methylation with other screening methods | 1 year
  Correlation coefficient of DNA methylation with high-risk HPV and TCT results

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China